CLINICAL TRIAL: NCT01807546
Title: A Phase II Study of Oral Rigosertib in Patients With Relapsed or Metastatic, Platinum-resistant, Human Papillomavirus Positive or Negative Squamous Cell Carcinoma
Brief Title: Oral Rigosertib for Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 09-09; COMIRB 13-0116 (Other: University of Colorado School of Medicine)
Record Dates: First submitted 2013-03-04; First posted 2013-03-08 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Anal Squamous Cell Carcinoma; Lung Squamous Cell Carcinoma; Cervical Squamous Cell Carcinoma; Esophageal Squamous Cell Carcinoma; Skin Squamous Cell Carcinoma; Penile Squamous Cell Carcinoma
Keywords: Head and neck cancer; Platinum-resistant; Squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Anus Neoplasms; Esophageal Squamous Cell Carcinoma; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rigosertib (Experimental): Oral rigosertib capsules at a dose of 560 mg twice a day for 14 consecutive days of a 21-day cycle (2 weeks on, 1 week off regimen).
  Interventions: Drug: rigosertib

INTERVENTIONS:
Drug: rigosertib — Oral rigosertib capsules at a dose of 560 mg twice a day for 14 consecutive days of a 21-day cycle (2 weeks on, 1 week off regimen).
  Other Names: ON 01910.Na

SUMMARY:
The primary objective of this study is to determine if tumors in patients with papillomavirus (HPV) positive or negative squamous cell carcinoma (SCC) that no longer responds to standard therapy will decrease in size following treatment with the investigational drug, rigosertib sodium (ON 01910.Na). A secondary objective is to determine if treatment with rigosertib causes any side effects.

Rigosertib is an investigational drug, which means that it has not been approved by the U.S. Food and Drug Administration (FDA) to treat any diseases. We are studying rigosertib as a new anticancer drug. Tests that we have done in the laboratory suggest that rigosertib works by blocking cell division in cancer cells and causing them to die.

DETAILED DESCRIPTION:
This will be a multicenter, Phase II study to evaluate the safety and efficacy of oral rigosertib in patients with relapsed or metastatic squamous cell carinoma (SCC) who previously received platinum-based chemotherapy and/or chemo-radiation therapy.

Only patients with head and neck squamous cell carinoma (HNSCC), non-small cell lung SCC, skin SCC, cervical SCC, penile SCC, anal SCC or esophageal SCC will be enrolled in the study.

Patients will be administered rigosertib capsules at a dose of 560 mg BID on days 1 to 14 of a 21-day cycle. Patients will be enrolled in 2 cohorts based on HPV test results:

* Cohort 1 will include up to 40 patients with human papillomavirus (HPV)-positive SCC, of which approximately 30 patients will have HNSCC, and approximately 10 patients with SCC of another origin (eg, cervix, anal, penile);
* Cohort 2 will include up to 40 patients with HPV-negative SCC, of which approximately 30 patients will have HNSCC, and approximately 10 patients with SCC of another origin (eg, lung, skin, esophageal).

Patients will be evaluated for progression after completing 3 cycles of therapy and every 3 cycles thereafter. Patients with stable disease (SD) or better, based on revised Response Criteria in Solid Tumors (mRECIST) 1.1, will receive repeated cycles of treatment on a 21-day cycle schedule until disease progression, development of unacceptable toxicity, or withdrawal of consent. Patients with progressive disease (PD) but who, in the opinion of the Investigator, appear to be deriving clinical benefit, may continue on study with a planned disease reassessment after one further cycle of therapy. Should the patient have SD or PR at this reassessment, s/he may continue on study, with subsequent reassessments every 3 cycles.

Following discontinuation of rigosertib treatment, patients' mortality status will be assessed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed SCC; only patients with HNSCC, non-small cell lung SCC, skin SCC, cervical SCC, penile SCC, anal SCC, or esophageal SCC;
2. For patients with HNSCC only, HPV status must be assessed by in situ hybridization (ISH) and/or p16 immunohistochemistry (IHC) according to local standards;
3. For patients with HNSCC only, HPV status must be assessed by in situ hybridization (ISH) and/or p16 immunohistochemistry (IHC) according to local standards. For all other patients with SCC originating in tissues other than the head and neck, attempts should be made to obtain HPV status;
4. Incurable, non-resectable, locally-advanced/relapsed and/or distant metastatic disease after no more than 3 prior treatment regimens, one of which must be platinum-based chemotherapy;
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤2;
6. Life expectancy of at least 3 months;
7. Measurable disease according to RECIST version 1.1;
8. Ability to swallow entire capsules;
9. Adequate hematologic function;
10. Adequate hepatic function;
11. Adequate renal function;
12. Adequate contraceptive regimens for female and male patients;
13. Female patients with reproductive potential must have a negative urine or serum pregnancy test;
14. Ability to understand the nature of the study and any hazards of study participation, to communicate satisfactorily with the Investigator, and to follow the requirements of the entire protocol;
15. Willingness to adhere to the prohibitions and restrictions specified in this protocol;
16. The patient must sign an informed consent form (ICF).

Exclusion Criteria:

1. Chemotherapy or any potentially myelosuppressive treatment within 3 weeks prior to enrollment (6 weeks are required for nitrosoureas or mitomycin C);
2. Radiotherapy to >25% of the hematopoietic active bone marrow within 4 weeks prior to enrollment;
3. Systemic administration of corticosteroids within the past 4 weeks prior to enrollment;
4. Prior therapy with a phosphatidylinositol 3-kinase (PI3K), Akt or mammalian target of rapamycin (mTOR) inhibitor;
5. Any other investigational agent or chemotherapy, radiotherapy, or immunotherapy within 4 weeks of enrollment;
6. Major surgery within 3 weeks of enrollment or major surgery without full recovery;
7. Residual clinical signs and symptoms which have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) version 4 Grade 1 severity level or below before enrollment, except for alopecia, stable residual neuropathy, and residual hand/foot syndrome;
8. Known brain metastases, except for those that have been removed or irradiated and have no current clinical impact at the time of enrollment; a computed tomography (CT) scan or magnetic resonance imaging (MRI) of the brain should be obtained in patients with symptoms suggestive of brain metastases;
9. Ascites requiring active medical management, including paracentesis;
10. Serum sodium less than 130 mEq/L or conditions that may predispose patients to hyponatremia (eg, previous syndrome of inappropriate antidiuretic hormone hypersecretion [syndrome of inappropriate antidiuretic hormone secretion (SIADH)], chronic diuretic use, etc.);
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, bleeding, symptomatic congestive heart failure, unstable angina pectoris, and cardiac arrhythmia;
12. Uncontrolled hypertension, defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥110 mmHg;
13. New onset of seizures within 3 months prior to enrollment, or poorly controlled seizures;
14. Psychiatric illness/social situations that would limit the patient's ability to tolerate and/or comply with study requirements;
15. History of allergic reactions attributed to compounds of similar chemical or biologic composition to rigosertib;
16. Female patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Baseline to 9 weeks after start of rigosertib treatment and every 9 weeks thereafter, up to 2 years.
  Outcome is defined as the number of patients with Complete Response (CR) or Partial Response (PR) per revised Response Evaluation Criteria In Solid Tumors (RECIST 1.1). Complete response (CR) is defined as disappearance of all target lesions. Partial Response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Overall survival (OS) | Date of signing ICF to date of death, or date last known to be alive up to 2 years after discontinuation of rigosertib treatment.
  At the time of analysis, the outcome measure will be number of days between the date the patient is enrolled in the study and the date the patient dies or date the patient is last known to be alive, up to 2 years following discontinuation of rigosertib treatment.
Progression free survival (PFS), | 9 weeks, 18 weeks, and 27 weeks and every 9 weeks thereafter, up to 2 years after patient enrolled in the study.
  At the time of analysis, the outcome measure will be number of days between the date the patient is enrolled in the study and the date that progressive disease (PD) is documented per revised Response Evaluation Criteria In Solid Tumors (RECIST 1.1).
Concentration of rigosertib in plasma | Cycle 1 Day 1, Cycle 1 Day 14 and Cycle 2 Day 14 at 0, 0.5, 1, 1.5, 2, and 6 hours after the first dose of the day.
  The concentration (expressed as microgram rigosertib per mL plasma and/or nanogram rigosertib per mL plasma) of rigosertib in plasma will be determined by a validated high performance liquid chromatography (HPLC) method.
Levels of Biomarkers | Baseline ( study before drug administration) and Cycle 1, Day 14.
  Genetic and protein profiling will be conducted in blood (collected at Baseline before study drug administration) and in core biopsy or fine needle aspirate tumor samples (collected at Baseline before study drug administration and at Cycle 1 Day 14).
Number of Adverse Events | From signing of Informed Consent Form until 30 days after last dose of study drug.
  All Adverse Events reported by the patient or observed by the Investigator or study site personnel will be recorded. An adverse event is defined as any unfavorable or unintended sign, symptom, or disease that appears or worsens in a patient during the period of observation in a clinical study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurman, MD, Study Director — Traws Pharma, Inc.
Locations (13):
- United States (13):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Stanford Cancer Institute, Stanford, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Denver VA Medical Center-ECHCS, Denver, Colorado
  - University of Michigan Health System, Ann Arbor, Michigan
  - Veterans Administration New Jersey Health Care System, East Orange, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University, James Cancer Hospital, Columbus, Ohio
  - University of Pennslvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Blue Ridge Cancer Care, Salem, Virginia

REFERENCES:
- [Background] Anderson RT, Keysar SB, Bowles DW, Glogowska MJ, Astling DP, Morton JJ, Le P, Umpierrez A, Eagles-Soukup J, Gan GN, Vogler BW, Sehrt D, Takimoto SM, Aisner DL, Wilhelm F, Frederick BA, Varella-Garcia M, Tan AC, Jimeno A. The dual pathway inhibitor rigosertib is effective in direct patient tumor xenografts of head and neck squamous cell carcinomas. Mol Cancer Ther. 2013 Oct;12(10):1994-2005. doi: 10.1158/1535-7163.MCT-13-0206. Epub 2013 Jul 19. PMID 23873848
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.